CLINICAL TRIAL: NCT04588441
Title: Aerosolized Inhaled Adenosine Treatment in Patients With Acute Respiratory Distress Syndrome (ARDS) Caused by COVID-19 (The ARCTIC Trial)
Brief Title: The ARCTIC Trial: Aerosolized Inhaled Adenosine Treatment in Patients With Acute Respiratory Distress Syndrome (ARDS) Caused by COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started due to need for additional preclinical work requested by FDA>
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202002127; OCR39505 (Other: UF OnCore)
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Distress
Keywords: COVID-19; ARDS; Adenosine
MeSH Terms: conditions — Acute Lung Injury; COVID-19 | interventions — Adenosine

STUDY DESIGN:
Intervention Model Description: Testing will be applied to patients with deteriorating pulmonary function and who are newly intubated (within 24 hours) with rising oxygen requirements.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adenosine (Experimental): Treatment consists of 9 mg adenosine in 5ml normal saline (NS) administered over 5-10 min via an Aerogen™ nebulizer
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Adenosine will be given like an inhaled asthma medication two times daily for one week (7 days). Treatment consists of 9 mg adenosine in 5ml normal saline (NS) administered over 5-10 min via an Aerogen™ nebulizer.
  Other Names: Aerogen

SUMMARY:
This is a phase II study to test adenosine efficacy for down-regulation of the overwhelming inflammation of COVID-19 in the lungs as reflected by clinical recovery of lung function; resolution of clinically relevant markers of lung function, and resolution of systemic markers of inflammation and coagulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) male and female patients with diagnosed COVID-19 respiratory infection, verified by culture/swab RNA. Impending ARDS respiratory collapse with progressive increasing oxygen requirements, and in line with sub-study as defined below.
* Patients intubated within the prior 24 hours.
* Hemodynamically stable (not requiring vasopressors or catecholamine agents to support systemic blood pressure; no existing shock defined as BP < 100 mmHg systolic).
* In-place continuous arterial line for blood sampling.

Exclusion Criteria:

* Younger than 18 years old.
* Prisoners
* Pregnant women.
* Unable to obtain next of kin consent.
* End-stage cardiac disease with COVID-19.
* Non COVID-related causes of ARDS/respiratory failure, septic shock, or post trauma shock, respiratory failure after blood transfusion or surgery.
* Unstable asthma or history of frequent/poorly controlled asthmatic attacks.
* Not expected to live more than 6 months due to underlying condition such as cancer.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improved COVID-19 symptoms | Day 50
  Improved COVID-19 symptoms measured by alive v. mortality, not hospitalized, or free of respiratory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Spiess, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No